CLINICAL TRIAL: NCT05360173
Title: Explore the Effectiveness of Acupressure on Reducing Pain and Improving Gastrointestinal Function of Patients After Laparoscopic Surgery
Brief Title: The Effectiveness of Acupressure on Reducing Pain and Improving Gastrointestinal Function After Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Li Chen, Adjunct Supervisor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMR-111-166
Record Dates: First submitted 2022-04-21; First posted 2022-05-04 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Pain
Keywords: Laparoscopic surgery; post-operative pain; acupressure; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: These two groups will be given true acupressure and sham acupressure twice daily. The participant will be observation the postoperative pain and postoperative recovery.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group not only have the routine treatment, but have acupressure when they back to the ward with the following 3 days . The effectiveness evaluation was carried out by the same researcher before and after intervention. There are three assessments in this study: primary outcome including postoperative pain and bowel movement. The short-form McGill Pain Questionnaire is used to measure the quality of pain, Visual Analog Scale is used to the pain intensity and stethoscope is used to listen to the bowel sound. The study, also, will be recorded postoperative exhaust time, the postoperative date of Indwelling drainage tube and postoperative length of stay.
  Interventions: Behavioral: acupressure
- Control group (Sham Comparator): The control group will have the same treatment and the evaluation, except received sham acupoint.
  Interventions: Behavioral: sham acupressure

INTERVENTIONS:
Behavioral: acupressure — The researcher use thumb and put about 3 kilogram on four acupoints where locating on the patient's arm and leg.
  Arms: Experimental group
Behavioral: sham acupressure — The researcher use thumb and put about 3 kilogram on four acupoints where locating at about 3 cm next to the acupoint on the patient's arm and leg.
  Arms: Control group

SUMMARY:
The purpose of the study is to explore the effect if acupressure reducing pain after laparoscopic surgery. The study is designed as an experimental research with repeat measurement design. The patients who are eligible for laparoscopic for general surgery and colorectal surgery in a medical center in the central part of Taiwan. The intervention of the research starts from the first date of postoperative day and the patient has the postoperative pain. The participant will be randomized into experimental group and control group. These two groups will be given true acupressure and sham acupressure twice daily. The participant will be observation the postoperative pain and postoperative recovery.

DETAILED DESCRIPTION:
Laparoscopic is increasing in this decade. The surgical trauma caused postoperative pain which cannot be avoid. It is the significant challenge and the thorny issue of the healthcare providers, also, be discussed for many decades. Several clinical researches have been verified acupuncture and related method have been as adjuvant efficacy treatment for decreasing postoperative pain. Acupressure is the method of the thumb put acupoint, and therapeutic effectiveness is similar to acupuncture. Acupressure is allowed to a nurse work independently due to noninvasive treatment. However, the less of the clinical studies explore the efficacy of acupressure reducing the postoperative pain after laparoscopic. The result of the research will provide the efficacy of reducing postoperative laparoscopic pain and wish to improve the quality of care.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic surgery on the organ of liver, gastric, small intestine, colon under general anaethesia
* the American Society of Anesthesiologists (ASA) :I - III
* above 20 years old
* the state of consciousness is alert
* Chinese or Taiwanese speaker

Exclusion Criteria:

* surgical procedure: resection, low anterior resection, Roux-en-Y Gastric Bypass and Whipple procedure (pancreaticoduodenectomy)
* postoperative length of hospital stay less than 3 days
* patient have pregnant, maternity, breastfeeding, chronic pain history, coagulation disorder or skin injury on the acupoints.
* drug abuse, alcoholism
* Patient-controlled analgesia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-06-16 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | 3 days
  Visual Analog Scale (VAS) of pain is used to measure the pain intensity. The scale of 0 = no pain and 10 = the worst pain, is a 10 cm scale marked in cm. The higher scores means the worse outcome.
The quality of postoperative pain | 3 days
  The short-form McGill Pain Questionnaire (SF-MPQ) is used to measure the quality of pain. The Chinese version is used that consists of 16 descriptors (12 sensory; 4 affective) which rated 0 = none, 1 = mild, 2 = moderate or 3 = severe, and Present Pain Intensity (PPI) and a visual analogue scale (VAS). The higher score means the worse outcome.
medication consumption | 3 days
  The data is recorded from the patient chart about the drugs consumption after surgery. That is included opioid, non-steroidal anti-Inflammatory drugs, prokinetic agent and anti-flatulence drugs. The more medications are used mean the worse outcome.

SECONDARY OUTCOMES:
Times of exhaust air | 3 days
  The data is recorded by ask the patient whether they have exhaust air or not after intervention. If the patient has exhaust air after the intervention, means the good outcome.
recovery of bowel movement | 3 days
  The stethoscope is used to listen to the bowel sound, which will be measured by the researcher. The bowel sound increase means the good outcome.
Timing of first flatus | 3 days
  asking the patient the timing of the first flatus after surgery, time is the shorter the better
postoperative length of stay | Postoperative day to discharge (about 5-7 days)
  recording from the chart, time is the shorter the better